CLINICAL TRIAL: NCT02558868
Title: Second-Line Oxaliplatin and Irinotecan Versus Irinotecan Alone for Advanced Pancreatic Cancer Patients Progressed After First-line Gemcitabine and S-1: A Randomized Controlled Study
Brief Title: Second-Line Oxaliplatin and Irinotecan Versus Irinotecan Alone for Gemcitabine and S-1 Refractory Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, Director, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYMedOncoPAC02
Record Dates: First submitted 2015-09-07; First posted 2015-09-24 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxaliplatin + Irinotecan (Experimental): Irinotecan：160 mg/m2，iv 120 min，d1 q2w oxaliplatin: 85 mg/m2，iv 120 min，d1 q2w
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin
- Irinotecan (Active Comparator): Irinotecan：180 mg/m2，iv 120 min，d1 q2w
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan
Drug: Oxaliplatin
  Arms: Oxaliplatin + Irinotecan

SUMMARY:
This study is a randomized, open-label, controlled study that will compare the efficacy of oxaliplatin in combination with irinotecan to irinotecan alone as second-line treatment for patients with gemcitabine and S-1 refractory pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced pancreatic cancer who had experienced progression during first-line gemcitabine and S-1 were eligible for enrollment on this open-label, randomized study.
* Additional inclusion criteria were age 18 years or older
* Measurable reference cancer site(s) confirmed with computed tomography (CT) or magnetic resonance imaging (MRI)
* Karnofsky performance status (KPS) of at least 70%
* -Adequate renal function, adequate hepatic function, adequate bone marrow function

Exclusion Criteria:

* The presence of any severe concomitant disease that could interrupt the planned treatment; intractable pain
* Hypersensitivity to study drugs
* Serious cardiovascular disease (eg, unstable coronary artery disease or myocardial infarction within 4 weeks of study start)
* National Cancer Institute CommonToxicity Criteria grade 3 or 4 sensory or motor neuropathy
* Prior or concurrent malignancy (other than pancreatic cancer)
* Female, pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 years

SECONDARY OUTCOMES:
Progression Free Survival | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, Doctor, Principal Investigator — First Affiliated Hospital,Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Oettle H, Riess H, Stieler JM, Heil G, Schwaner I, Seraphin J, Gorner M, Molle M, Greten TF, Lakner V, Bischoff S, Sinn M, Dorken B, Pelzer U. Second-line oxaliplatin, folinic acid, and fluorouracil versus folinic acid and fluorouracil alone for gemcitabine-refractory pancreatic cancer: outcomes from the CONKO-003 trial. J Clin Oncol. 2014 Aug 10;32(23):2423-9. doi: 10.1200/JCO.2013.53.6995. Epub 2014 Jun 30. PMID 24982456